CLINICAL TRIAL: NCT06676345
Title: Mechanical Complications of Acute Myocardial Infarction: a Multicenter Prospective Observational Study
Brief Title: Mechanical Complications of Acute Myocardial Infarction: a Multicenter Prospective Study
Acronym: CAUTION 2
Status: Recruiting | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: IT-VA:56/2024
Record Dates: First submitted 2024-11-01; First posted 2024-11-06 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Ventricular Septal Defect; Papillary Muscle Rupture; Cardiac Rupture; Pseudoaneurysm
MeSH Terms: conditions — Heart Septal Defects, Ventricular; Heart Rupture; Aneurysm, False | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with post-infarction mechanical complications: All the patients diagnosed with post-infarction mechanical complications, independently from the treatment assigned (surgical, percutaneous or conservative)
  Interventions: Procedure: Surgical treatment; Procedure: Percutaneous treatment

INTERVENTIONS:
Procedure: Surgical treatment — Surgical repair of post-infarction mechanical complications (e.g. sutureless or sutured repair for LVFWR, David or Daggett technique for VSR, mitral valve repair or replacement for PMR)
Procedure: Percutaneous treatment — Percutaneous approach for the management of post-infarction mechanical complications (e.g. percutaneous closure with device for VSR, Mitraclip for PMR, PIFIT for LVFWR)

SUMMARY:
In 2019, the international study titled "CAUTION Study - 1" (MeChanical complicAtions of acUte myocardial infarcTion: an InternatiOnal multiceNter cohort study), a retrospective multicenter study, was launched and registered on ClinicalTrials.gov (Identifier: NCT03848429). This study highlighted the outcomes of surgical treatment of post-infarction mechanical complications in patients operated between 2000 and 2019. Several scientific publications have resulted from this registry, which involved 27 international centers and recruited about 800 patients. However, retrospective studies are inherently limited by factors such as selection bias and a high number of missing data, affecting data interpretation and consistency of results. Moreover, most registries report only data about surgical patients or, in rare situations, about patients treated percutaneously. To overcome these limitations, a prospective study has been designed to collect more precise and focused data and achieve results that better reflect the current clinical practice, including all the patients diagnosed with post-infarction mechanical complications, independently from the treatment assigned.

"CAUTION Study - 2" is, therefore, a prospective, multicenter cohort study with the primary aim of analyzing the outcomes of surgical, percutaneous and conservative treatment of post-infarction mechanical complications in the contemporary era.

DETAILED DESCRIPTION:
In Western countries, cardiovascular diseases are the leading cause of death among people over 65 years old. Acute myocardial infarction represents the most frequent cardiovascular event among the heart diseases. In recent years, with the spread of percutaneous coronary reperfusion techniques, there has been a reduction in the incidence of mechanical complications of acute myocardial infarction. However, mortality in patients who develop one of these complications remains high, with mechanical complications representing a relevant cause of death in patients with acute coronary syndrome after cardiogenic shock and arrhythmia.

The acute mechanical complications of myocardial infarction include ventricular free-wall rupture (VFWR), ventricular pseudo-aneurysm, acute mitral regurgitation due to papillary muscle rupture (PMR), and ventricular septal rupture (VSR). Numerous surgical techniques and management protocols have been proposed to address these complications, but the most effective ones and those associated with better outcomes remain unclear. Recently, percutaneous treatment techniques have also been proposed in this setting (particularly for VSD and PMR), especially for high-risk surgical patients or those considered inoperable, though the safety and efficacy of these approaches remain uncertain.

In 2019, the international study titled "CAUTION Study - 1" (MeChanical complicAtions of acUte myocardial infarcTion: an InternatiOnal multiceNter cohort study), a retrospective multicenter study, was launched and registered on ClinicalTrials.gov (Identifier: NCT03848429). This study highlighted the outcomes of surgical treatment of post-infarction mechanical complications in patients operated between 2000 and 2019. Several scientific publications have resulted from this registry, which involved 27 international centers and recruited about 800 patients. However, retrospective studies are inherently limited by factors such as selection bias and a high number of missing data, affecting data interpretation and consistency of results. Moreover, most registries report only data about surgical patients or, in rare situations, about patients treated percutaneously. To overcome these limitations, a prospective study has been designed to collect more precise and focused data and achieve results that better reflect the current clinical practice, including all the patients diagnosed with post-infarction mechanical complications, independently from the treatment assigned.

"CAUTION Study - 2" is, therefore, a prospective, multicenter cohort study with the primary aim of analyzing the outcomes of surgical, percutaneous and conservative treatment of post-infarction mechanical complications in the contemporary era.

Data on patients undergoing surgical, percutaneous or conservative treatment for post-infarction mechanical complications will be prospectively collected from participating Departments of Cardiac Surgery and Cardiology from January 1st, 2025, to December 31st, 2027. According to the "CAUTION Study 1", each center treats an average of 5-10 patients per year for mechanical complications of acute myocardial infarction. Therefore, considering that at least 50 centers will participate in this study, the goal is to recruit approximately 800 patients, making this the largest prospective study on these conditions. Clinically relevant patient data will be anonymized and entered by individual centers into a dedicated data collection platform (e.g., RedCap). The accuracy of data entry will be verified by the study's promoting center, which will also handle the statistical analysis and data processing.

For every participating center, it is expected that approximately 10-15 patients will be enrolled. For each patient, demographic and clinical data such as age, gender, diagnosis, key laboratory tests, diagnostic procedures performed during hospitalization, associated diseases, description of the surgical intervention or percutaneous procedure, post-operative complications, and in-hospital outcomes will be recorded. Analysis of quality of life, the need for new hospitalizations or re-interventions, and long-term survival of recruited patients will be conducted during the annual follow-up visit, which all patients usually undergo, or through access to the regional or national electronic health record.

Patient enrollment will take place after they have reviewed the information sheet "Informed Consent to Participate in the Study: CAUTION Study 2" and have provided their consent.

ELIGIBILITY:
Inclusion Criteria:

* all the patients diagnosed with post-infarction mechanical complications, independently from the treatment assigned

Exclusion Criteria:

* patients with cardiac rupture not acute myocardial infarction related

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients diagnosed with post-infarction mechanical complications
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
In-hospital mortality | from enrollment to the end of hospitalization (up to 30 days)
  Mortality during the hospitalization for the management of post-infarction mechanical complication

SECONDARY OUTCOMES:
Long-term survival | from enrollment to the end of follow-up (5 years from diagnosis)
  Survival at 5 years from the diagnosis of post-infarction mechanical complication

CONTACTS AND LOCATIONS:
Locations (1):
- ASST dei Sette Laghi, Varese, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ronco D, Matteucci M, Kowalewski M, De Bonis M, Formica F, Jiritano F, Fina D, Folliguet T, Bonaros N, Russo CF, Sponga S, Vendramin I, De Vincentiis C, Ranucci M, Suwalski P, Falcetta G, Fischlein T, Troise G, Villa E, Dato GA, Carrozzini M, Serraino GF, Shah SH, Scrofani R, Fiore A, Kalisnik JM, D'Alessandro S, Lodo V, Kowalowka AR, Deja MA, Almobayedh S, Massimi G, Thielmann M, Meyns B, Khouqeer FA, Al-Attar N, Pozzi M, Obadia JF, Boeken U, Kalampokas N, Fino C, Simon C, Naito S, Beghi C, Lorusso R. Surgical Treatment of Postinfarction Ventricular Septal Rupture. JAMA Netw Open. 2021 Oct 1;4(10):e2128309. doi: 10.1001/jamanetworkopen.2021.28309. PMID 34668946
- [Background] Matteucci M, Ronco D, Kowalewski M, Massimi G, De Bonis M, Formica F, Jiritano F, Folliguet T, Bonaros N, Sponga S, Suwalski P, De Martino A, Fischlein T, Troise G, Dato GA, Serraino FG, Shah SH, Scrofani R, Kalisnik JM, Colli A, Russo CF, Ranucci M, Pettinari M, Kowalowka A, Thielmann M, Meyns B, Khouqeer F, Obadia JF, Boeken U, Simon C, Naito S, Musazzi A, Lorusso R. Long-term survival after surgical treatment for post-infarction mechanical complications: results from the Caution study. Eur Heart J Qual Care Clin Outcomes. 2024 Dec 19;10(8):737-749. doi: 10.1093/ehjqcco/qcae010. PMID 38327179
- [Background] Matteucci M, Kowalewski M, De Bonis M, Formica F, Jiritano F, Fina D, Meani P, Folliguet T, Bonaros N, Sponga S, Suwalski P, De Martino A, Fischlein T, Troise G, Dato GA, Serraino GF, Shah SH, Scrofani R, Antona C, Fiore A, Kalisnik JM, D'Alessandro S, Villa E, Lodo V, Colli A, Aldobayyan I, Massimi G, Trumello C, Beghi C, Lorusso R. Surgical Treatment of Post-Infarction Left Ventricular Free-Wall Rupture: A Multicenter Study. Ann Thorac Surg. 2021 Oct;112(4):1186-1192. doi: 10.1016/j.athoracsur.2020.11.019. Epub 2020 Dec 9. PMID 33307071